CLINICAL TRIAL: NCT06880679
Title: Use of Point-of-Care Ultrasound (POCUS) for the Diagnosis of Acute Chest Syndrome in Patients With Sickle Cell Disease
Brief Title: Ultrasound Acute Chest Syndrome Sickle Cell Disease
Acronym: POCUS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Seethal Jacob, MD, MS, Associate Professor of Pediatrics, Indiana University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PHO-IIR-POCUS
Record Dates: First submitted 2025-02-17; First posted 2025-03-18 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2025-04

CONDITIONS: Acute Chest Syndrome; Sickle Cell Disease
Keywords: Sickle Cell Disease; Sickle Cell Anemia; Acute Chest Syndrome; POCUS; Ultrasound
MeSH Terms: conditions — Acute Chest Syndrome; Anemia, Sickle Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Ultrasound (Experimental): Ultrasound days 1, 3, and 5 of hospitalization
  Interventions: Device: Point of Care Ultrasound

INTERVENTIONS:
Device: Point of Care Ultrasound — Point of Care Ultrasound during hospitalization

SUMMARY:
Feasibility and reliability of ultrasound in the inpatient hematology setting.

DETAILED DESCRIPTION:
Acute chest syndrome (ACS) is a complication of sickle cell disease where individuals have symptoms of fever, low oxygen levels or difficulty breathing in the setting of a new lung finding on chest x-ray. Chest x-ray is a useful tool to identify it but has some side effects. The investigators think ultrasound will be an equally feasible, reliable tool and minimize some of the side effects associated with chest x-ray. Ultrasound is a non-invasive was to obtain an image that does not require radiation.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 0-25 years old
2. Diagnosis: Patients with a documented diagnosis of sickle cell disease (any genotype)
3. Disposition: Hospitalized for a SCD-related complication (e.g. VOC)

Exclusion Criteria:

1. Patient is considered hemodynamically unstable to undergo consent and study procedures
2. Already has diagnosis of ACS prior to admission to inpatient unit
3. POCUS operator not available

Max Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-04-08 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Participation rate | Up to 5 days
  Percentage of patients who are approached for study who agree to be on study
Retention rate | Up to 5 days
  Percentage of patients who remain on study
Duration of exam | Up to 5 days
  Time taken to complete POCUS examination
Acceptability of POCUS by the medical team (physicians and nursing) | Up to 5 days
  Acceptability measured using a 5-point Likert Scale (Strongly Agree to Strongly Disagree) regarding use of POCUS in inpatient setting.

SECONDARY OUTCOMES:
Reliability of point of care ultrasound (POCUS) compared to standard of care (Chest X-ray) | Up to 5 days
  A positive screening of acute chest syndrome by POCUS is identification of either a lung consolidation or focal B-lines. POCUS findings will be compared to standard of care (Chest X-ray) findings to see if findings concur.

CONTACTS AND LOCATIONS:
Overall Officials: Seethal Jacob, MD, Principal Investigator — Indiana University
Locations (1):
- Indiana University, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No